CLINICAL TRIAL: NCT05874687
Title: Tricuspid Annular Plane Systolic Excursion to Predict Arterial Hypotension Caused by Spinal Anesthesia in Caesarean Section
Acronym: CESERAN TAPSE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aydin Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, MEDİCİNE DOCTOR, Aydin Maternity and Child Health Hospital
Other Study IDs: 2023-
Record Dates: First submitted 2023-05-11; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hypotension
Keywords: Tricuspid Annuler Plane Systolic Excursion; Hypotension-; Ceserean section; Spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Coal Tar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: hypotension +,: hypotension +: hypotension defined as a decreased SAB greater than 20% of baseline, a decreased MAP below 90 mmHg, or a MAP of 65 mmHg
  Interventions: Drug: hypotension + treat
- 2:hypotension -: hypotension -:none hypotension (hypotension defined as a decreased SAB greater than 20% of baseline, a decreased MAP below 90 mmHg, or a MAP of 65 mmHg)

INTERVENTIONS:
Drug: hypotension + treat — Heart Rate and Mean Arterial Pressure (MAP) will be recorded throughout the procedure (every 2 minutes for the first 15 minutes). Ephedrine (in 6 mg increments) will be used as well as the isotonic balanced crystalloid solution to treat hypotension defined as a decreased SAB greater than 20% of baseline, a decreased MAP below 90 mmHg, or a MAP of 65 mmHg (250 mL bolus). The Ephedrine dose will be recorded. Bradycardia, which is defined as a heart rate less than 50 beats per minute, will be treated with intravenous Atropine (0.5 mg).
  Groups: 1: hypotension +,

SUMMARY:
This cross-sectional blinded study was planned to be conducted in Aydın Gynecology and Pediatrics Hospital between June 2023 and September 2023. The study was designed for adult pregnant female cases between the ages of 20 and 35. Patients with Class II American Society of Anesthesiologists (ASA) physical status, scheduled for elective cesarean section under subarachnoid block and who gave informed consent were planned to be included in the study.

Patients with emergencies and uncontrolled systemic comorbidities (e.g., cardiovascular, respiratory or renal) and patients with expected massive intraoperative loss (i.e., placenta accreta or placenta previa) are planned to be excluded from the study. Also, cases receiving intravenous fluid preload will be excluded.

DETAILED DESCRIPTION:
This cross-sectional blinded study was planned to be conducted in Aydın Gynecology and Pediatrics Hospital between June 2023 and September 2023. The study was designed for adult pregnant female cases between the ages of 20 and 35. Patients with Class II American Society of Anesthesiologists (ASA) physical status, scheduled for elective cesarean section under subarachnoid block and who gave informed consent were planned to be included in the study.

Patients with emergencies and uncontrolled systemic comorbidities (e.g., cardiovascular, respiratory or renal) and patients with expected massive intraoperative loss (i.e., placenta accreta or placenta previa) are planned to be excluded from the study. Also, cases receiving intravenous fluid preload will be excluded.

Echocardiography The same observer will perform TTE on all patients in the left lateral decubitus position with an echocardiography device. The values of all parameters will be determined by taking the average values of three cardiac cycle measurements. Measurement methods will be used in accordance with the guidelines of the American Society of Echocardiography. M-Mode, 2D (2D) images, color, pulse and continuous wave Doppler and tissue Doppler measurements will be taken from all subjects who are suitable for standard Echocardiography. LV Ejection Fraction (EF) measurements will be evaluated in the parasternal long axis view.

FAC and TAPSE will be used to evaluate Right Ventricular (RV) systolic functions. Tricuspid E and A Wave Velocity and E/A Ratio will be measured to evaluate the diastolic function of the RV. TAPSE, echocardiography device and TTE will be used for all patients by the same observer. Echocardiography will be performed in the left lateral supine position. TAPSE will be calculated in an apical 4-chamber view by placing an M-mode cursor across the Tricuspid Ring and measuring the amount of longitudinal movement at peak systole and the values will be recorded by averaging the five cardiac cycle measurements.

Patients will be visualized in the supine position through the subxiphoid window of the Inferior Vena Cava (IVC). The cursor will be placed 1 cm distal to the hepatic vein IVC entry point and the IVC diameter will be monitored for 30 seconds in M-Mode. And the measurement will be made from the region where the diameter of the inferior vena cava is in inspiration (IVCins) and expiration (IVCexp) while the patient is breathing normally. The Inferior Vena Cava Collapse Index (IVC-CI) will be calculated by using the formula IVC-CI = (IVCexp - IVCins) / IVCexp.

Spinal Anesthesia Following the echocardiographic measurements, spinal anesthesia will be administered with 2.1 mL of hyperbaric Bupivacaine 5% to the L 4-5 or L 3-4 intervertebral spaces with a 25-gauge spinal needle in the sitting position. All patients will then be simultaneously loaded with a Ringer's Lactate solution (10 mL/kg over 15 minutes). Surgery will be started when the sensory block reaches the T6 level.

Heart Rate and Mean Arterial Pressure (MAP) will be recorded throughout the procedure (every 2 minutes for the first 15 minutes). Ephedrine (in 6 mg increments) will be used as well as the isotonic balanced crystalloid solution to treat hypotension defined as a decreased SAB greater than 20% of baseline, a decreased MAP below 90 mmHg, or a MAP of 65 mmHg (250 mL bolus). The Ephedrine dose will be recorded. Bradycardia, which is defined as a heart rate less than 50 beats per minute, will be treated with intravenous Atropine (0.5 mg).

The present study aimed to determine the predictive values of IVCCI and IJVCI in determining PSAH. The secondary purpose was to compare these two predictive values.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 2
2. 37-42 gestational-week single pregnancies
3. Being between the ages of 20-35
4. BMI between 20-35

Exclusion Criteria:

1. Non-sinus rhythm
2. ASA III and above
3. Known heart disease
4. Multiple pregnancy
5. Expected massive intraoperative loss (i.e., placenta accreta or placenta previa)
6. Severe pulmonary hypertension, wall motion disorder, severe valve disease, hypertrophic or dilated cardiomyopathy in echocardiography
7. A TAPSE value of 1.7 cm or less

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Due to the cesarean section, only female patients will be included in the study.
Study Population: The study was designed for adult pregnant female cases between the ages of 20 and 35. Patients with Class II American Society of Anesthesiologists (ASA) physical status, scheduled for elective cesarean section under subarachnoid block and who gave informed consent were planned to be included in the study
Sampling Method: Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
ceserenan tapse | 3 months
  The primary outcome measure was the development of hypotension after spinal anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydin Maternity and Child Health Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided